CLINICAL TRIAL: NCT03518437
Title: Coronary Atherosclerosis Disease Early Identification and Risk Stratification by Noninvasive Imaging :A Cohort Study of China
Brief Title: Coronary Atherosclerosis Disease Early Identification and Risk Stratification by Noninvasive Imaging
Acronym: Creation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Bin Lu, Director of radiology department, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CIFuwaiHospital-1
Record Dates: First submitted 2016-09-19; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; CT; MACE
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — bio-markers of coronary artery disease
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigator prospectively enroll 30,000 outpatients who were suspected of coronary artery disease (CAD) and underwent cardiac computed tomography angiography (CTA). The endpoint was major adverse cardiac events (MACE).The investigator aim to evaluate the prognostic value of CTA, risk factors and bio-markers for MACE.

DETAILED DESCRIPTION:
The investigator prospectively enroll 30,000 outpatients who were suspected of coronary artery disease (CAD) and underwent cardiac computed tomography (CT). Cardiac CT was assessed for coronary artery calcification score (CACS) and the extent, the location, the stenosis severity, and the composition of the plaque in CTA. The base line information was recorded, including risk factors, drugs, bio-markers, and psychological. The endpoint was MACE, defined as composite cardiac death, nonfatal myocardial infarction (MI).we aim to evaluate the prognostic value of CTA, risk factors and bio-markers for major adverse cardiac events (MACE).

ELIGIBILITY:
Inclusion Criteria:

1. suspected of coronary heart disease, coronary CTA has been completed.
2. age > 18 years old.
3. have biochemical test results.
4. signed informed consent.

Exclusion Criteria:

1. malignant tumor, severe liver and kidney diseases.
2. combination of cardiomyopathy, valvular disease, congenital heart disease, a variety of reasons the left cardiac insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We prospectively enroll 30,000 outpatients who were suspected of coronary artery disease (CAD) and underwent cardiac computed tomography (CT)
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events | 3 years
  cardiac death, myocardial infarction (Cardiac death was defined as death due to acute myocardial infarction, ventricular arrhythmias, refractory heart failure or cardiogenic shock. The investigator reviewed all available data to determine whether a cardiac etiology was the immediate cause of death and categorized cardiac deaths into sudden cardiac death and nonsudden cardiac death. Sudden cardiac death was defined by published criteria . myocardial infarction was defined based on the criteria of typical chest pain, elevated cardiac enzyme levels and typical alterations of the electrocardiogram. )

CONTACTS AND LOCATIONS:
Overall Officials: bin lu, M.D., Study Chair — Chinese Academy of Medical Sciences
Locations (1):
- Binlu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] SCOT-HEART investigators. CT coronary angiography in patients with suspected angina due to coronary heart disease (SCOT-HEART): an open-label, parallel-group, multicentre trial. Lancet. 2015 Jun 13;385(9985):2383-91. doi: 10.1016/S0140-6736(15)60291-4. Epub 2015 Mar 15. PMID 25788230
- [Result] Hou ZH, Lu B, Gao Y, Jiang SL, Wang Y, Li W, Budoff MJ. Prognostic value of coronary CT angiography and calcium score for major adverse cardiac events in outpatients. JACC Cardiovasc Imaging. 2012 Oct;5(10):990-9. doi: 10.1016/j.jcmg.2012.06.006. PMID 23058065
- [Result] Shah R, Foldyna B, Hoffmann U. Outcomes of anatomical vs. functional testing for coronary artery disease : Lessons from the PROMISE trial. Herz. 2016 Aug;41(5):384-90. doi: 10.1007/s00059-016-4451-3. PMID 27333988
- [Result] Min JK, Dunning A, Lin FY, Achenbach S, Al-Mallah M, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Cheng V, Chinnaiyan K, Chow BJ, Delago A, Hadamitzky M, Hausleiter J, Kaufmann P, Maffei E, Raff G, Shaw LJ, Villines T, Berman DS; CONFIRM Investigators. Age- and sex-related differences in all-cause mortality risk based on coronary computed tomography angiography findings results from the International Multicenter CONFIRM (Coronary CT Angiography Evaluation for Clinical Outcomes: An International Multicenter Registry) of 23,854 patients without known coronary artery disease. J Am Coll Cardiol. 2011 Aug 16;58(8):849-60. doi: 10.1016/j.jacc.2011.02.074. PMID 21835321